CLINICAL TRIAL: NCT05300984
Title: Evaluation of the Anti-aging Efficacy of a Novel Cosmetic Product
Brief Title: Evaluation of the Anti-aging Efficacy of a Novel Skin Health Product
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amazentis SA (Industry)
Collaborators: proDERM GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 22.01.AMZ; 22.0052-23 (Other: proderm GmbH)
Record Dates: First submitted 2022-03-19; First posted 2022-03-29 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Skin Aging
Keywords: Mitochondria, Aging
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Split face/arm design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental)
  Interventions: Other: Topical Placebo Cream; Other: Topical Cream with 0.5% Active
- Group 2 (Experimental)
  Interventions: Other: Topical Placebo Cream; Other: Topical Cream with 1% Active

INTERVENTIONS:
Other: Topical Placebo Cream — cosmetic cream to be applied topically on face and forearms twice/daily using split/face design
Other: Topical Cream with 0.5% Active — cosmetic cream to be applied topically on face and forearms twice/daily using split/face design
  Arms: Group 1
Other: Topical Cream with 1% Active — cosmetic cream to be applied topically on face and forearms twice/daily using split/face design
  Arms: Group 2

SUMMARY:
The aim of this study is to investigate the effect of cosmetic products with two different concentrations of the active on skin aging and in acting on the mitochondrial health of skin in comparison to a placebo product.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent to participate in the study
* Willingness to actively participate in the study and to come to the scheduled visits
* Female
* From 50 to 75 years of age
* Visible wrinkle in the face (grade 3 to 6 according to proderm scale) see Appendix 2
* Healthy skin in the test areas
* Vaccination of tetanus within the last 10 years (for biopsy sub group)

Exclusion Criteria:

* Female subjects: Pregnancy or lactation
* Drug addicts, alcoholics
* AIDS, HIV-positive or infectious hepatitis
* Conditions which exclude a participation or might influence the test reaction/evaluation
* Participation or being in the waiting period after participation in cosmetic and/or pharmaceutical studies pertaining to the test area
* Cancer not being diagnosed as cured and requiring chemotherapy, irradiation and/or hormonal treatment within the last 2 years
* Diabetes mellitus (type 1 and 2)
* One of the following illnesses with reduced physical capability/fitness: asthma (symptom-free allergic asthma is not an exclusion criterion), hypertension, cardiovascular diseases
* Documented allergies to cosmetic products and/or ingredients, skin care and/or skin cleansing products
* Intolerability against adhesive dressing (e.g. acrylate)
* Active skin disease at the test area
* Regular use of tanning beds
* Wounds, moles, tattoos, scars, irritated skin, excessive hair growth, etc. at the test area that could influence the investigation
* Any topical medication at the test area within the last 3 days prior to the start of the study
* Medical treatment for wrinkle reduction (e.g. peeling with vitamin A or fruit acids) on the face within the last 2 weeks prior to the start of the study
* Systemic therapy with immuno-suppressive drugs (e.g. corticosteroids) and/or antihistamines (e.g. antiallergics) within the last 7 days prior to the start of the study
* Systemic therapy with anti-phlogistic agents or analgetics (e.g. diclophenac), except for minor pain relief medicine like paracetamol within the last 3 days prior to the start of the study
* Therapy with antibiotics within the last 2 weeks prior to the start of the study
* Regular medication with anti-coagulating drugs like Aspirin®, Macumar®, etc. (e.g. for thrombosis prophylaxis) within up to 15 days prior to the taking of the biopsies
* Past cosmetic surgery procedure in the test area (e.g. laser, facelift)
* History of complications at wound healing (e.g. keloids, hypertrophic scars or contracture scar)

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 48 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
Change from baseline in skin mitochondrial health and biological age (assessed on skin biopsies) after 8 weeks | 8 weeks
Change from baseline in skin barrier function (assessed on transepidermal waterloss by Tewameter [g/(m²h)]) after 8-weeks | 8 weeks

SECONDARY OUTCOMES:
Change from baseline in skin barrier function (assessed on transepidermal waterloss by Tewameter [g/(m²h)]) after 2-weeks | 2-weeks
Change from baseline in skin hydration (assessed on skin capacitance by Corneometer [a.u.]) after 2 and 8 weeks | 8 weeks
Change from baseline in pigmentation (assessed on skin color by Spectrophotometer) after 2 and 8 weeks | 8 weeks
Change from baseline in skin firmness by Cutometer [mm] after 2 and 8 weeks | 8 weeks
Change from baseline in skin elasticity by Cutometer after 2 and 8 weeks | 8 weeks
Change from baseline in skin layer thickness and undulation index of DEJ (assessed on Line field confocal Optical Coherence Tomography Image analysis) after 8 weeks for both groups or after 2 and 8 weeks | 8 weeks
Change from baseline for wrinkles and fine lines (assessed on Colorface Image analysis) after 2 and 8 weeks | 8 weeks
Subjective Evaluation of product traits assessed via questionnaire after 2 and 8 weeks | 2 and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. med. Klaus-Peter Wilhelm, Dermatologist, MD, Study Chair — proDERM GmbH; Dr. rer. nat. Sabrina Laing, MD, Principal Investigator — proDERM GmbH
Locations (1):
- proderm GmbH, Schenefeld, Germany

IPD SHARING:
Plan to Share IPD: No